CLINICAL TRIAL: NCT01347424
Title: Evaluating Endostatin Plus TC Regimen in Secondary Malignant Neoplasm of Liver Using Contrast Enhancement Ultrasonography
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XIANSHENG
Record Dates: First submitted 2011-04-27; First posted 2011-05-04 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2010-11

CONDITIONS: Non Small Cell Lung Cancer; Nasopharyngeal Cancer; Liver Metastasis
Keywords: NSCLC; NPC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Nasopharyngeal Neoplasms | interventions — Paclitaxel; Carboplatin; Endostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test group (Experimental)
  Interventions: Drug: Paclitaxel , carboplatin, endostatin
- control group (Active Comparator)
  Interventions: Drug: Paclitaxel and Carboplatin

INTERVENTIONS:
Drug: Paclitaxel , carboplatin, endostatin — PTX：175mg/m2，D1, q3w CBP：AUC5，D1, q3w endostatin：7.5 mg/m2 iv 3-4h， d1～15，q3w
  Arms: Test group
Drug: Paclitaxel and Carboplatin — PTX：175mg/m2，D1, q3w CBP：AUC5，D1, q3w
  Arms: control group

SUMMARY:
Contrast enhancement ultrasonography（CEUS）could be used to evaluate the blood flow perfusion liver cancer. In this clinical trial, CEUS was used to evaluated the changes of blood flow perfusion of Secondary Malignant Neoplasm of Liver after treated with endostatin plus paclitaxel and carboplatin regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of nasopharyngeal carcinoma or NSCLC
* With an evaluable secondary malignant neoplasm of Liver, diameter≥2cm
* Without transcatheter arterial chemoembolization (TACE) treatment
* Performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) Scale.
* Estimated life expectancy of at least 3 months
* Patient compliance and geographic proximity that allow adequate follow-up.
* Adequate organ function including the following: Bone marrow: absolute neutrophil count (ANC) >or= 1.5x10^9/L, platelets >or= 100x10^9/L, hemoglobin >or= 9g/dL. Hepatic: bilirubin <1.5 x ULN, alkaline phosphatase, aspartate transaminase (AST) and alanine transaminase (ALT) < 2.5 x ULN (alkaline phosphatase, AST, ALT < 5 x ULN is acceptable if liver has tumor involvement). Renal: calculated creatinine clearance > 45 ml/min.
* Men or women of at least 18 years of age.
* Signed informed consent from patient.

Exclusion Criteria:

* Women who are pregnant or in lactation
* Systemic treatment for another cancer within the year prior to study entry
* Known hypersensitivity to any of the study drugs or to drugs with similar chemical structures
* Use of investigational agents within 28 days of the Baseline visit, or participating simultaneously in any other clinical studies
* Severe co-morbidity of any type that may interfere with assessment of the patient for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-05 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
The changes of blood flow perfusion in secondary malignant neoplasm of liver | 12months

SECONDARY OUTCOMES:
Comparing the difference of OS(Overall Survival) and ORR(Objective Response Rate) according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria in the two different arms. | 12 months
Number of Participants with Adverse Events in the two different arms | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Principal Investigator — Cancer Center of Sun Yat-Sen University (CCSU)
Locations (1):
- SunYat-senU, Guangzhou, Guangdong, China